| ID | #: |
|----|----|

## PARENT/GUARDIAN CONSENT FORM

# NU-HOME New Ulm-Healthy Home Offerings via the Mealtime Environment

You are invited to be in a research study to test a program about family meals. You were selected as a possible participant because you have a 7-10 year old child. Also, you make most of the meals your family eats at home. We ask that you read this form and ask any questions before agreeing to be in the study.

This study is being conducted by Jayne A. Fulkerson, PhD from the University of Minnesota in collaboration with Rebecca Lindberg, MPH from the Minneapolis Heart Institute Foundation and Abbey Sidebottom, MPH, PhD from Allina Health.

## **Background Information**

The purpose of the NU-HOME study is to test a program that encourages families to eat meals together and eat healthy foods. The program also encourages families to be physical active together.

#### **Procedures:**

If you agree to be in this study, we would ask you to do the following things:

- 1) Participate in data collection.
  - a. We will collect data from families 3 times over the course of a year and a half. At each data collection visit, you and your child will have your height and weight measured. You and your child will also answer questions about physical activity, the foods you eat, and cooking and eating at home with your family. You and your child will also participate in two interviews about the food your child has eaten in the past 24 hours. Your child will also wear a physical activity tracker for 7 days to measure physical activity.
  - b. There will be 2 additional short data collection visits during the year and a half. At each of these data collection visits, <u>your child's</u> height and weight will be measured. Also, your child will answer questions about physical activity.
- 2) Allow you and your family to be randomly assigned to be in one of two groups.
  - a. If your family is randomly assigned to the NU-HOME group, your family will participate in a program to increase the frequency of family meals and healthful foods at meals. The program will focus on meal planning, cooking skills and recipes, nutrition education, and how to be more physically active. The format will be useful for parents and fun for children. We will ask that you and your family attend seven monthly sessions (two hours long) starting in the fall. Sessions will be held at a location in your community.

OR

| ID #: |
|-------|

b. If your family is randomly assigned to the other group, your family will participate in a similar program about family meals and healthful food at meals. However, this program will start after the research study is over.

Both you and your 7-10 year old child must agree to participate for your family to be in the study. Although only your 7-10 year old child complete surveys and height and weight measurement, the rest of your household is invited to attend the NU-HOME program sessions.

## Risks and Benefits of being in the Study

The study has minimal risks. You may feel uncomfortable having your height and weight measured. Trained study staff will take measurements in a private area and will not share the results with you or any other family member unless you give us permission. You may feel uncomfortable answering questions about your eating and physical activity habits. You are free to skip any question you prefer not to answer without any penalty. Your family may have some conflict about changing the food offerings or television limits in your home. The choice to change your home environment is up to you.

There are no direct benefits to participation. We will provide dinner, and childcare and transportation will be provided if needed.

## Compensation:

Your family will receive gift cards for completing each family data collection visit. At each family visit, you will receive \$25 for height and weight measurement and for answering the survey questions that day. Over the following two weeks, you will receive an additional \$25 gift card for completing one additional phone interview about the food your child had to eat the previous day and returning the physical activity tracker your child wore for 7 days. You will receive a third \$25 gift card for completing the snack and evening meal screener surveys. Thus, if you complete all of the planned data collection at each data collection period, your family will receive \$75 each time (total of \$225 in gift cards per family if you complete all data collection at each of the 3 data collection time points).

# Confidentiality:

We will use electronic devices (ipads, phones, computers) for data collection using a secure REDCap database and a secure web interface. The records from this study will be stored securely and kept private. A secure username and password will be required to access the records and only researchers on the study team will have access. However, your study records may be reviewed by University regulatory staff if they have appropriate oversight approval. We will not include any information in publications or presentation that will make it possible to identify you. To these extents, confidentiality is not absolute. Study data will be encrypted according to current University policy for protection of confidentiality.

The following information is not limited by confidentiality and may be released as governed by law: 1) information about a child being maltreated or neglected 2) information about an individual's plan to seriously harm him/herself 3) information about an individual's plan to seriously harm another person.

| | ID #: |
|---|---|
| Voluntary Nature of the Study: Participation in this study is voluntary. Your decision whether or not affect your current or future relations with the University of Minneso Minneapolis Heart Institute Foundation. If you decide to participate, answer any question or withdraw at any time without affecting those | ta, Allina Health, or the you are free to not |
| Contacts and Questions: If you have questions about research appointments, the study, reseconcerns you may ask questions now or if you have questions later to contact Dr. Fulkerson at 308 Harvard Street, Minneapolis, MN 58 fulke001@umn.edu. | , you are encouraged |
| To share feedback privately, about your research experience include the study, call the Research Subjects' Advocate Line (612) 625-165 online at <a href="https://www.irb.umn.edu/report.html">www.irb.umn.edu/report.html</a> . You may also contact the H Protection Program in writing at D528 Mayo, 420 Delaware St. Sou Minnesota 55455. | 50 or give feedback<br>luman Research |
| You will be given a copy of this information to keep for your re | ecords. |
| Statement of Consent: I have read the above information. I have asked questions and have consent to participate in the study. | e received answers. I |
| Signature of participant: | Date: |
| Signature of person explaining study: | Date: |
| Consent for photographs I agree to allow my family to be photographed as part of the NU-HC The photographs may be used in NU-HOME presentations and ma presentations, and for other research purposes. I understand that in materials my family's name will not be associated with photo image | terials, in professional any presentations or |
| Statement of Consent: I have read the above information. I have asked guestions and have | e received answers. |
| □Yes | |

Signature of participant:\_\_\_\_\_ Date: \_\_\_\_\_

☐ No

| Research in the Future | |
|---|---|
| would be interested in participating in addition you be interested in letting us contact you in | NU-HOME families in the future to see if they onal measurements or a future study. Would the future? Giving us permission to contact of future studies. Please check one of the lines |
| Statement of Consent: I have read the above information. I have as | ked questions and have received answers. |
| I give my consent for NU-HOME additional research opportunitie | E staff to <b>contact me in the future</b> about es. |
| I <b>do not</b> want NU-HOME staff to research opportunities. | o contact me in the future about additional |
| Signature of participant: | Date: |

ID #: \_\_\_\_\_